CLINICAL TRIAL: NCT00185705
Title: Randomized, Placebo Controlled, Double Blind Trial of Telmisartan in Hypertensive, Obese Adolescents
Brief Title: Treatment of Insulin Resistance in Hypertensive, Obese Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigator moved to different university
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carolyn Chi, Principle Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Telmisartan adolescents
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Hypertension; Insulin Resistance; Dyslipidemia
Keywords: Insulin resistance; obesity; hypertension; adolescents; telmisartan; lifestyle intervention
MeSH Terms: conditions — Hypertension; Insulin Resistance; Dyslipidemias; Obesity | interventions — Telmisartan

INTERVENTIONS:
Drug: Telmisartan

SUMMARY:
In this study, we propose using telmisartan, an angiotensin II receptor antagonist with PPAR-gamma modulating activity, for a 12-week period to decrease blood pressure and insulin levels in obese, hypertensive children. Telmisartan is currently approved for treatment of adult hypertension. Recent adult studies, however, have shown telmisartan as an effective medication for lowering insulin levels and improving insulin sensitivity. We will enroll 30 obese adolescents, ages 10 to 18 years, and randomly assign half of the group to receive telmisartan and the other half to receive placebo (sugar-pill). We will obtain fasting glucose and insulin levels, as well as other markers for insulin sensitivity and cholesterol panel, at the beginning of the study, at each clinic visit in 4-week intervals, and at the end of the study. We will obtain an imaging study (computed tomography, CT scan) on 10 randomly selected study patients (5 from each group) to examine the distribution of fat tissue before and after treatment. Studies suggest that fat tissue in the subcutaneous tissue is less harmful that fat tissues surrounding internal organs, such as the liver. We will also provide nutritional handouts and exercise recommendations to each participant as a life-style intervention. Each participant will be given a diary to record his or her diet and exercise activities throughout the study.

DETAILED DESCRIPTION:
Hypothesis: This pilot study will provide data essential for designing a larger trial to test the hypothesis that telmisartan treatment of obese children with insulin resistance and hypertension will result in improved insulin levels and systolic blood pressure. Secondary outcome measures will include the effects of telmisartan on total cholesterol, triglyceride, HDL and LDL levels, body mass index (BMI), and body fat distribution.

Specific Aims for to Test Hypothesis:

Aim #1: Determine the change in insulin sensitivity in adolescents with obesity and hyperinsulinemia before and after treatment with telmisartan. We hypothesize a significant increase in insulin sensitivity following medical treatment. We will measure fasting insulin and glucose levels for calculation of the homeostasis model assessment (HOMA) [29, 30]. Furthermore, we will calculate parameters of insulin production and insulin resistance from simultaneous measurements of glucose, insulin, and C-peptide levels during an oral glucose tolerance test (OGTT). We will check IGF BP-1 (insulin-like growth factor 1 binding protein) level as an indirect measurement of insulin resistance. Due to the risks associated with glucose clamps and continuous insulin infusion, we will not use this procedure in our study.

Aim #2: Determine the change in systolic blood pressure in adolescents with obesity and hypertension before and after treatment with telmisartan. We hypothesize a significant decrease in systolic blood pressure following medical treatment. Subjects will have blood pressure checked at each clinic visit.

Aim #3: Evaluate changes in lipid profile and body mass index as secondary outcome measures with telmisartan treatment. Subjects will have weight, height, and fasting lipid panel checked at each clinic visit.

Aim #4: Characterize fat distribution before and after telmisartan treatment. A subset of study participants will undergo magnetic resonance imaging (MRI) to characterize and separate abdominal adipose tissue into its subcutaneous and visceral components. A one-slice MRI will be obtained at 2 time-points during the study (weeks 0 and 12).

Aim #5: Determine the feasibility of using telmisartan for the treatment of hyperinsulinemia and hypertension in obese adolescents. Study results will provide necessary data to calculate the power needed for a multi-center, randomized, placebo-controlled trial of telmisartan.

ELIGIBILITY:
Inclusion Criteria:

Ages between 10.00 and 17.99 years

Body mass index (BMI) ≥ 95th percentile for age and gender using the CDC data

SBP ≥ 95th percentile for age, gender, and height using the fourth report from the National High Blood Pressure Education Program (NHBPEP) guidelines.

Fasting plasma insulin concentration ≥ 20 U/mL will be required for study entry. This insulin concentration is commonly used for defining insulin resistance.

Exclusion Criteria:

Subjects will be excluded from the study if they have known diabetes as defined by the American Diabetes Association criteria, prior drug therapy to treat diabetes or insulin resistance, recent glucocorticoid therapy within 3 months of the screening visit, current drug therapy to treat hypertension, elevated creatinine (> 1.2mg/dL), elevated liver enzymes (ALT > 80), history or current alcohol ingestion, existing pregnancy or high-risk of becoming pregnant, other serious medical condition that the investigator determines may put the subject at undue risk if enrolled in the study, or taking medications with potential drug-drug interactions (anticoagulant, digoxin, diuretics).

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
This pilot study will provide data essential for designing a larger trial to test the hypothesis that telmisartan treatment of obese children with insulin resistance and hypertension will result in improved insulin levels and systolic blood pressure.

SECONDARY OUTCOMES:
Secondary outcome measures will include the effects of telmisartan on total cholesterol, triglyceride, HDL and LDL levels, body mass index (BMI), and body fat distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn H Chi, MD, Principal Investigator — Stanford Medical Center
Locations (1):
- Stanford Medical Center, Stanford, California, United States

REFERENCES:
- [Background] Berenson GS. Childhood risk factors predict adult risk associated with subclinical cardiovascular disease. The Bogalusa Heart Study. Am J Cardiol. 2002 Nov 21;90(10C):3L-7L. doi: 10.1016/s0002-9149(02)02953-3. PMID 12459418
- [Background] Duncan GE, Li SM, Zhou XH. Prevalence and trends of a metabolic syndrome phenotype among u.s. Adolescents, 1999-2000. Diabetes Care. 2004 Oct;27(10):2438-43. doi: 10.2337/diacare.27.10.2438. PMID 15451913
- [Background] de Ferranti SD, Gauvreau K, Ludwig DS, Neufeld EJ, Newburger JW, Rifai N. Prevalence of the metabolic syndrome in American adolescents: findings from the Third National Health and Nutrition Examination Survey. Circulation. 2004 Oct 19;110(16):2494-7. doi: 10.1161/01.CIR.0000145117.40114.C7. Epub 2004 Oct 11. PMID 15477412
- [Background] Ferrannini E, Haffner SM, Mitchell BD, Stern MP. Hyperinsulinaemia: the key feature of a cardiovascular and metabolic syndrome. Diabetologia. 1991 Jun;34(6):416-22. doi: 10.1007/BF00403180. PMID 1884900
- [Background] Freedman DS, Khan LK, Dietz WH, Srinivasan SR, Berenson GS. Relationship of childhood obesity to coronary heart disease risk factors in adulthood: the Bogalusa Heart Study. Pediatrics. 2001 Sep;108(3):712-8. doi: 10.1542/peds.108.3.712. PMID 11533341
- [Background] Hardin DS, Hebert JD, Bayden T, Dehart M, Mazur L. Treatment of childhood syndrome X. Pediatrics. 1997 Aug;100(2):E5. doi: 10.1542/peds.100.2.e5. PMID 9233976
- [Background] Kaplan F, Al-Majali K, Betteridge DJ. PPARS, insulin resistance and type 2 diabetes. J Cardiovasc Risk. 2001 Aug;8(4):211-7. doi: 10.1177/174182670100800405. PMID 11550999
- [Background] Kurtz TW, Pravenec M. Antidiabetic mechanisms of angiotensin-converting enzyme inhibitors and angiotensin II receptor antagonists: beyond the renin-angiotensin system. J Hypertens. 2004 Dec;22(12):2253-61. doi: 10.1097/00004872-200412000-00003. PMID 15614015
- [Background] Owens S, Gutin B, Barbeau P, Litaker M, Allison J, Humphries M, Okuyama T, Le NA. Visceral adipose tissue and markers of the insulin resistance syndrome in obese black and white teenagers. Obes Res. 2000 Jul;8(4):287-93. doi: 10.1038/oby.2000.34. PMID 10933304
- [Background] Sinaiko AR, Steinberger J, Moran A, Prineas RJ, Jacobs DR Jr. Relation of insulin resistance to blood pressure in childhood. J Hypertens. 2002 Mar;20(3):509-17. doi: 10.1097/00004872-200203000-00027. PMID 11875319
- [Background] Sorof JM, Lai D, Turner J, Poffenbarger T, Portman RJ. Overweight, ethnicity, and the prevalence of hypertension in school-aged children. Pediatrics. 2004 Mar;113(3 Pt 1):475-82. doi: 10.1542/peds.113.3.475. PMID 14993537
- [Background] Steinberger J, Daniels SR; American Heart Association Atherosclerosis, Hypertension, and Obesity in the Young Committee (Council on Cardiovascular Disease in the Young); American Heart Association Diabetes Committee (Council on Nutrition, Physical Activity, and Metabolism). Obesity, insulin resistance, diabetes, and cardiovascular risk in children: an American Heart Association scientific statement from the Atherosclerosis, Hypertension, and Obesity in the Young Committee (Council on Cardiovascular Disease in the Young) and the Diabetes Committee (Council on Nutrition, Physical Activity, and Metabolism). Circulation. 2003 Mar 18;107(10):1448-53. doi: 10.1161/01.cir.0000060923.07573.f2. No abstract available. PMID 12642369
- [Background] Teo K, Yusuf S, Sleight P, Anderson C, Mookadam F, Ramos B, Hilbrich L, Pogue J, Schumacher H; ONTARGET/TRANSCEND Investigators. Rationale, design, and baseline characteristics of 2 large, simple, randomized trials evaluating telmisartan, ramipril, and their combination in high-risk patients: the Ongoing Telmisartan Alone and in Combination with Ramipril Global Endpoint Trial/Telmisartan Randomized Assessment Study in ACE Intolerant Subjects with Cardiovascular Disease (ONTARGET/TRANSCEND) trials. Am Heart J. 2004 Jul;148(1):52-61. doi: 10.1016/j.ahj.2004.03.020. PMID 15215792
- [Background] Yamagishi S, Takeuchi M. Telmisartan is a promising cardiometabolic sartan due to its unique PPAR-gamma-inducing property. Med Hypotheses. 2005;64(3):476-8. doi: 10.1016/j.mehy.2004.09.015. PMID 15617852
- [Background] Benson SC, Pershadsingh HA, Ho CI, Chittiboyina A, Desai P, Pravenec M, Qi N, Wang J, Avery MA, Kurtz TW. Identification of telmisartan as a unique angiotensin II receptor antagonist with selective PPARgamma-modulating activity. Hypertension. 2004 May;43(5):993-1002. doi: 10.1161/01.HYP.0000123072.34629.57. Epub 2004 Mar 8. PMID 15007034
- [Background] Derosa G, Ragonesi PD, Mugellini A, Ciccarelli L, Fogari R. Effects of telmisartan compared with eprosartan on blood pressure control, glucose metabolism and lipid profile in hypertensive, type 2 diabetic patients: a randomized, double-blind, placebo-controlled 12-month study. Hypertens Res. 2004 Jul;27(7):457-64. doi: 10.1291/hypres.27.457. PMID 15302981